CLINICAL TRIAL: NCT06285162
Title: Analgesia Nociception Index and Autonomic Nervous System Exploration During Continuous Renal Replacement Therapy in Intensive Care Patients.
Brief Title: Analgesia Nociception Index to Explore Autonomic Nervous System in Patients With Continuous Renal Replacement Therapy
Acronym: UFANI
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL23_1372; 2024-A00294-43 (Other: ID-RCB)
Record Dates: First submitted 2024-02-22; First posted 2024-02-29 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Critically Ill; Renal Replacement Therapy
Keywords: Analgesia Nociception Index; R-R interval; autonomic nervous system; haemodynamic; fluid removal
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Critically ill patients with continuous renal replacement therapy.: The patients will be followed during the first 6 hours of the initiation of a net ultrafiltration (2-3 milliliters/kilograms/hour) with continuous monitoring (R-R interval, ANI, cardiac index, invasive arterial pressure, central venous pressure, peripheral perfusion index), and perfusion monitoring every 6 hours (arterial lactate, central venous oxygen saturation, capillary refill time, mottling score). Such a fluid removal strategy is part of an institutional protocol or an ongoing clinical trial.
  In addition to the usual monitoring, the PhysioDoloris monitor will be connected to the patient's scope. The ANI and its parameters will be recorded continuously throughout the study.

SUMMARY:
The Analgesia Nociception Index (ANI) reflects the balance between sympathetic and parasympathetic tone. It is based on a specific interpretation of the R-R interval variation. During fluid removal by net ultrafiltration in patients with fluid overload and continuous renal replacement therapy, some data suggest that haemodynamic variation could be induced by the autonomic nervous system. The study aims to investigate ANI variations in this context and their association with the haemodynamic variations observed.

ELIGIBILITY:
Inclusion Criteria:

* Continuous renal replacement therapy in intensive care unit
* Initiation of net ultrafiltration according to the protocol of the department or to EARLYDRY study (NCT 05817539) (3 criteria required):

  * Fluid overload > 5% or peripheral oedema
  * Noradrenaline equivalent <0.5μg/kg/min
  * No peripheral hypoperfusion
* Invasive blood pressure monitoring
* Central venous line in superior vena cava territory
* Regular sinus rhythm
* Patient awake or Richmond Agitation and Sedation Scale > -3

Exclusion Criteria:

* Ongoing administration of inotropes
* Ongoing administration of beta blockers
* Current administration of alpha-2 agonists
* History of dysautonomia
* Pregnant or breast-feeding woman
* Mechanical circulatory assistance
* Opposition to participate
* Adults under legal protection
* Persons deprived of their liberty by judicial or administrative decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients with continuous renal replacement therapy, fluid overload and haemodynamically stable.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2026-01-09 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Percentage of changes in ANI. | 6 hours after initiation of net ultrafiltration
  Relative changes in ANI (averaged over 4 minutes (percentage)) between Hour 0 and Hour 6 of initiation of net ultrafiltration.

CONTACTS AND LOCATIONS:
Overall Officials: Martin RUSTE, MD, Principal Investigator — Département d'anesthésie-réanimation, Hôpital cardiologique Louis Pradel, HCL
Locations (1):
- Département d'anesthésie-réanimation Hôpital cardiologique Louis Pradel, Bron, France